CLINICAL TRIAL: NCT00610506
Title: A Pilot Study -- An Open-Label, Rater-blinded, Flexible-dose, 8-week Trial of Escitalopram (Lexapro®) In Patients With Major Depression With Atypical Features.
Brief Title: Escitalopram (Lexapro®) In Patients With Major Depression With Atypical Features
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 7842; IRB#7842
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2008-01

CONDITIONS: Atypical Depression
Keywords: Atypical Depression
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Lexapro
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram will be started at 10 mg per day and augmented weekly in 10 mg per day increments, the maximum dose being 20 mg per day. The dose will be titrated upward or downward based on clinical response and tolerability.
  Other Names: Escitalopram (Lexapro)

SUMMARY:
Aims of Study:

The aims of this study are 1) to examine the clinical utility of escitalopram in patients with major depression with atypical features; 2) to evaluate the tolerability of escitalopram in major depression with atypical features.

Study hypothesis and objectives. This study is proposed as an open-label study to gather pilot data to examine whether escitalopram has clinical utility in the treatment of major depression with atypical features. Because of the exploratory nature of the design, no specific study hypotheses can be generated regarding efficacy of the drug. Our primary hypothesis is that the effect size of escitalopram in atypical depression will be similar to the effect size of escitalopram in major depression, its FDA approved indication.

DETAILED DESCRIPTION:
Based on treatment outcome, longitudinal course, biologic and physiologic data, and family histories (Rabkin et al., 1996), the American Psychiatric Association's Diagnostic and Statistical Manual, Fourth Edition (DSM-IV) (American Psychiatric Association, 1994) added atypical features as a parenthetical modifier of major depression and dysthymia. Several recent reports suggest that DSM-IV criteria for depression with atypical features identify a group distinguishable by a cluster of symptoms, age of onset and course of illness. The symptom constellation consists of depressed mood, along with hyperphagia, weight gain, increased fatigue and rejection sensitivity. Some authors have distinguished two subtypes of atypical depression. One subtype has an early onset (i.e., before age 20 years) and a chronic course (i.e., no spontaneous well-being since onset greater than 2 months) (early/chronic atypical) are no more likely to benefit from tricyclic antidepressant than from placebo (Stewart et al., 2002), but do respond to a monoamine oxidase inhibitor, and do not have increased left hemisphere perceptual processing (Stewart et al., 2003). In contrast, the other subtype reports either later onset or a less chronic course of illness (late/nonchronic atypical) respond robustly to tricyclic antidepressant (Stewart et al., 2002), and show evidence of increased left hemispheric processing (Stewart et al., 2003).

The role of the newer medications in the treatment of depressed patients with atypical features remains to be elucidated. One study compared outcome between phenelzine and fluoxetine, reporting no difference, but risk of a type II error was large (Pande et al. 1996). A second study limited to depressed patients with atypical features compared fluoxetine, imipramine, and placebo, finding both drugs effective for about half the patients and both superior to placebo, but not different from each other (McGrath et al. 2000). A 12-week study comparing moclobemide and sertraline in the treatment of outpatients with atypical depression found both drugs to produce comparable improvement (Sogaard et al, 1999). Falkai (1999) asserts the efficacy of mirtazapine for depression with atypical features without any data, and Rye et al. (1998) reported on a single case of apparently late onset atypical depression responding to bupropion. A placebo controlled study failed to show any benefit for mianserin for atypical depression (McGrath et al, 1985). Finally, an unmarketed drug, gepirone, has been demonstrated to be effective for depression with atypical features but no comparison was made with other antidepressant medications (McGrath et al., 1994).

Escitalopram has been approved for the treatment of major depression and Generalized Anxiety Disorder. However whether escitalopram improved atypical depressive symptoms has not been investigated.

Aims of Study:

The aims of this study are 1) to examine the clinical utility of escitalopram in patients with major depression with atypical features; 2) to evaluate the tolerability of escitalopram in major depression with atypical features.

Study hypothesis and objectives. This study is proposed as an open-label study to gather pilot data to examine whether escitalopram has clinical utility in the treatment of major depression with atypical features. Because of the exploratory nature of the design, no specific study hypotheses can be generated regarding efficacy of the drug. Our primary hypothesis is that the effect size of escitalopram in atypical depression will be similar to the effect size of escitalopram in major depression, its FDA approved indication.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 65 years,
2. DSM-IV episode of Major Depression non-psychotic with atypical features.
3. ≥19 score on the 29-item HAM-D,
4. ability to give informed consent, if patients are of child-bearing potential
5. A minimum 2-week washout from existing psychotropics (5 weeks for fluoxetine).

Exclusion Criteria:

1. bipolar depression,
2. Any Axis I psychotic disorder
3. currently suicidal or suicide risk,
4. history of substance abuse in the previous 12 months,
5. history of hypersensitivity to escitalopram, or citalopram
6. serious or unstable medical disorders,
7. starting or terminating psychotherapy during the previous 12 weeks,
8. ECT treatment in the previous 3 months,
9. pregnancy or planning pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
changes in HAM-D-29 scores from baseline to end of treatment. | 8 weeks

SECONDARY OUTCOMES:
changes in 8-atypical items on the HAM-D-29, SDS and ESQ from baseline to end of treatment. Response will be defined as 50% or greater reduction in HAM-D-29 scores from baseline to end of treatment. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aswin A Patkar, M.D., Principal Investigator — Duke University
Locations (1):
- Dept Psychiatry, Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Pae CU, Masand PS, Peindl K, Mannelli P, Han C, Marks DM, Patkar AA. An open-label, rater-blinded, flexible-dose, 8-week trial of escitalopram in patients with major depressive disorder with atypical features. Prim Care Companion J Clin Psychiatry. 2008;10(3):205-10. doi: 10.4088/pcc.v10n0305. PMID 18615172